CLINICAL TRIAL: NCT00636831
Title: Prophylactic Antibiotic Use in Inguinal Hernioplasty: A Placebo-controlled, Double-blind Trial
Brief Title: Prophylactic Antibiotic Use in Hernioplasty
Acronym: RCT-herniation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon University (Other)
Responsible Party: Principal Investigator, Takero Mazaki, MD, PhD, Dr, Nihon University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Hikari-0701
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Inguinal Hernia
Keywords: Prophylactic; Antibiotic; Infection; Primary case
MeSH Terms: conditions — Hernia, Inguinal; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- cont (Placebo Comparator)
  Interventions: Drug: Antibiotic: cefazolin Sodium
- intervention (Active Comparator)
  Interventions: Drug: Antibiotic: cefazolin Sodium

INTERVENTIONS:
Drug: Antibiotic: cefazolin Sodium — 1g continuous IV at 30 minutes before starting operation

SUMMARY:
The purpose of this study is to determine whether prophylactic antibiotic use in inguinal hernioplasty are effective in prevention of infectious complication.

ELIGIBILITY:
Inclusion Criteria:

* Primary inguinal hernia
* Elective surgery
* Must be older than 20 years of age
* Must not have any serious complication

Exclusion Criteria:

* Incarceration
* Recurrence
* Drug allergy
* Diabetes mellitus
* Malignant diseases
* Serious heart diseases
* Psychological diseases
* Pregnancy
* Have been medicated with corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
infectious complication | two year

SECONDARY OUTCOMES:
Recurrence of inguinal hernia | two year

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon University School of Medicine, Department of Surgery, Tokyo, Japan